CLINICAL TRIAL: NCT02627144
Title: AVASTIN® First Line in Metastatic Renal Cancer
Brief Title: Bevacizumab in Metastatic Renal Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21519
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Renal Cell Cancer
Keywords: Metastatic renal cell carcinoma; Avastin; Bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Advanced and/or Metastatic RCC participants: Participants with mRCC who are being treated with bevacizumab at the recommended dose of 10 milligram per kilogram (mg/kg) of body weight once every 2 weeks as an intravenous infusion, in combination with interferon alpha-2a at the recommended starting dose of 9 million international units (MIU) 3 times a week until disease progression will be observed. No diagnostic or therapeutic interventions will be given other than used in normal daily routine.
  Interventions: Drug: Bevacizumab; Drug: Interferon alpha-2a

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered at the recommended dose of 10 mg/kg of body weight once every 2 weeks as an intravenous infusion until disease progression.
  Other Names: Avastin
Drug: Interferon alpha-2a — Interferon alpha-2a will be administered at the recommended starting dose of 9 MIU 3 times a week until disease progression.

SUMMARY:
This is a non-interventional, multicenter study to evaluate efficacy and safety of intravenous bevacizumab (Avastin) in combination with interferon alpha-2a immunotherapy for first-line treatment in participants with advanced and/or metastatic renal cell cancer (mRCC) in daily routine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced and/or metastatic renal cell cancer
* No contraindications for Avastin according to summary of product characteristics (SmPC)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced and/or metastatic renal cell cancer
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2008-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Schultze-Seemann W, Schulz H, Tschechne B, Hackl M. Bevacizumab plus IFN-alpha-2a in First-line Treatment of Patients With Advanced or Metastatic Renal Cell Carcinoma: A Prospective German Non-interventional Study. Anticancer Res. 2019 Feb;39(2):875-882. doi: 10.21873/anticanres.13188. PMID 30711970

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced and/or Metastatic RCC Participants: Participants with metastatic renal cell cancer (mRCC) who were treated with bevacizumab at the recommended dose of 10 milligram per kilogram (mg/kg) of body weight once every 2 weeks as an intravenous infusion, in combination with interferon alpha-2a at the recommended starting dose of 9 million international units (MIU) 3 times a week until disease progression were observed. No diagnostic or therapeutic interventions were given other than used in normal daily routine.
Period: Overall Study
Arm/Group | Advanced and/or Metastatic RCC Participants
Started | 365
Treated | 359
Completed | 0
Not Completed | 365
Not completed — Serious adverse event | 32
Not completed — Cancer progression | 171
Not completed — Death from cancer | 20
Not completed — Death from other cause | 8
Not completed — Refusal of treatment / poor cooperation | 38
Not completed — Administrative reasons | 65
Not completed — Lost to Follow-up | 8
Not completed — Enrolled, not treated | 6
Not completed — Other | 17

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who have received at least once one dose of bevacizumab.
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.1)
Sex/Gender, Customized [Number; unit: participants]
  Male | 242
  Female | 114
  Not available | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Tumor Response
Description: Tumor response was assessed as one of the following: Complete response (CR): disappearance of all target lesions and all pathological lymph nodes below 10 millimeter (mm). Partial response (PR): At least a 30 percent (%) decrease in the sum of diameters of target lesions. Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions.
Time Frame: Baseline until progression or intolerable toxicity, whichever occurred first, assessed up to 6 years
Population: Full analysis set (FAS) included all participants who received at least one dose of study medication and have at least one post dose efficacy assessment, following the intention-to-treat principle. 'Number of participants analyzed' indicate participants with non-missing tumor response data.
Measure: Number; unit: percentage of participants
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 338
percentage of participants
  CR | 5.3
  PR | 21.9
  SD | 39.1
  PD | 16.6
  Not Evaluable | 17.2

2. Primary Outcome: Percentage of Participants With Disease Control
Description: Disease control was defined as having achieved CR, PR, and/or SD during the course of the observation. CR: disappearance of all target lesions and all pathological lymph nodes below 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions.
Time Frame: Baseline until progression or intolerable toxicity, whichever occurred first, assessed up to 6 years
Population: FAS. 'Number of participants analyzed' indicate participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 338
percentage of participants | 66.3

3. Primary Outcome: Progression-free Survival (PFS) Time
Description: PFS time is defined as time between start of therapy and progression or death. Kaplan-Meier estimate was used for evaluation. PD: At least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm or persistence of non-target lesions.
Time Frame: Baseline until progression or intolerable toxicity or death, whichever occurred first, assessed up to 6 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 354
months | 10.2 [8.6 to 12.6]

4. Primary Outcome: Overall Survival (OS) Time
Description: OS time is defined as time between start of therapy and date of death. Kaplan-Meier estimate was used for evaluation.
Time Frame: Baseline until progression or intolerable toxicity or death, whichever occurred first, assessed up to 6 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 354
months | 28.7 [24.5 to 38.3]

5. Primary Outcome: Cumulative Dose of Immunotherapy (Interferon Alpha-2a) in Daily Routine
Time Frame: Up to 52 weeks
Population: FAS. Data were not analyzed for this outcome measure as therapy doses and pattern were not recorded numerically.
Arm/Group | Advanced and/or Metastatic RCC Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 6 years
Description: Safety set
Arm/Group | Advanced and/or Metastatic RCC Participants
Serious Adverse Events (participants affected / at risk) | 72/359
Other Adverse Events (participants affected / at risk) | 325/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced and/or Metastatic RCC Participants (N=359)
Cerebral haemorrhage (Nervous system disorders) | 4
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 3
Epilepsy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
General physical health deterioration (General disorders) | 6
Asthenia (General disorders) | 2
Death (General disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 6
Hypertensive crisis (Vascular disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Diverticulitis (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Confusional state (Psychiatric disorders) | 4
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Weight decreased (Investigations) | 2
Cerebral atrophy (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Orthostatic intolerance (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Senile dementia (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Impaired healing (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Angiodysplasia (Vascular disorders) | 1
Arterial thrombosis (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Rectal tenesmus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abscess intestinal (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aortic valve sclerosis (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Bladder tamponade (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Blood glucose abnormal (Investigations) | 1
Amaurosis (Eye disorders) | 1
Retinal exudates (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Sciatica (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced and/or Metastatic RCC Participants (N=359)
Anaemia (Blood and lymphatic system disorders) | 198
Leukopenia (Blood and lymphatic system disorders) | 150
Thrombocytopenia (Blood and lymphatic system disorders) | 118
Neutropenia (Blood and lymphatic system disorders) | 83
Influenza like illness (General disorders) | 146
Pyrexia (General disorders) | 116
Pain (General disorders) | 85
Fatigue (General disorders) | 42
Spinal pain (General disorders) | 18
Nausea (Gastrointestinal disorders) | 140
Diarrhoea (Gastrointestinal disorders) | 80
Vomiting (Gastrointestinal disorders) | 65
Hypertension (Vascular disorders) | 107
Proteinuria (Renal and urinary disorders) | 90
Back pain (Musculoskeletal and connective tissue disorders) | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 24
Peripheral sensory neuropathy (Nervous system disorders) | 44
Headache (Nervous system disorders) | 37
Dizziness (Nervous system disorders) | 21
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 54
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 34
Cardiac failure (Cardiac disorders) | 27
Weight decreased (Investigations) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.